CLINICAL TRIAL: NCT05170594
Title: A Prospective Study of Bevacizumab Combined With Fluzoparib, Bevacizumab Combined With Chemotherapy or Fluzoparib Monotherapy in the Treatment of Platinum-resistant Recurrent Ovarian Cancer
Brief Title: A Study of Bevacizumab Combined With Fluzoparib/Chemotherapy or Fluzoparib in the Treatment of Ovarian Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Shandong First Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MT-004
Record Dates: First submitted 2021-12-24; First posted 2021-12-28 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Ovarian Cancer
Keywords: platinum-resistant; recurrent ovarian cancer; Bevacizumab; Fluzoparib
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Bevacizumab; Drug Therapy; fluzoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bevacizumab combined with Fluzoparib (Experimental): Bevacizumab combined with Fluzoparib will be administered in patients with platinum-resistant recurrent ovarian cancer.
  Interventions: Drug: Bevacizumab; Drug: chemotherapy
- Bevacizumab combined with chemotherapy (Experimental): Bevacizumab combined with non-platinum chemotherapy will be administered in patients with platinum-resistant recurrent ovarian cancer.
  Interventions: Drug: Bevacizumab; Drug: chemotherapy
- Fluzoparib (Experimental): Fluzoparib monotherapy will be administered in patients with platinum-resistant recurrent ovarian cancer.
  Interventions: Drug: Fluzoparib

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab will be administered at 15mg/kg IV, every 3 weeks
  Other Names: Antiangiogenic drugs
  Arms: Bevacizumab combined with Fluzoparib; Bevacizumab combined with chemotherapy
Drug: chemotherapy — The non-platinum chemotherapy regimen will be determined by the investigator.
  Other Names: Non-platinum chemotherapy
  Arms: Bevacizumab combined with Fluzoparib; Bevacizumab combined with chemotherapy
Drug: Fluzoparib — Fluzoparib will be administered orally continuously at 150mg bid until disease progression and toxicity becomes intolerable
  Other Names: PARPi
  Arms: Fluzoparib

SUMMARY:
This study was designed to explore the safety and efficacy of Bevacizumab combined with Fluzoparib, Bevacizumab combined with chemotherapy or Fluzoparib monotherapy in patients with platinum-resistant recurrent ovarian cancer.

DETAILED DESCRIPTION:
This purpose of this study is to explore efficacy of Bevacizumab combined with Fluzoparib, Bevacizumab combined with chemotherapy or Fluzoparib monotherapy in patients with platinum-resistant recurrent ovarian cancer.Besides the efficacy,we focus on the safety and quality of life in the new treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, female;
2. Recurrent epithelial ovarian cancer, fallopian tube cancer, or primary peritoneal cancer proven to be platinum-resistant by histology or cytology;
3. ECOG score was 0-1;
4. Expected survival time > 12 weeks;
5. Normal or abnormal bone marrow, kidney, and liver function of the patient has no clinical significance, and the specific situation will be comprehensively determined by the investigator;
6. Patients not previously treated with PARPi or targeted drugs;
7. The patient has taken effective contraceptive measures within 14 days prior to screening and is willing to sign the notification until the last medication No pregnancy plan and voluntary use of effective contraceptive measures within the next 6 months;
8. The subject or his/her legal guardian can communicate well with the investigator, understand and comply with the requirements of this study, and understand and sign the informed consent.

Exclusion Criteria:

1. Known allergy to fluzopalil or study drug components;
2. Patients with any factors affecting oral administration (such as previous gastric or small bowel resection, or current atrophic gastritis, chronic intestinal disease, gastrointestinal bleeding, dysphagia, gastrointestinal obstruction, or diarrhea greater than grade 1, including those who have recovered but have not recovered);
3. Patients who underwent major surgery or gastrointestinal surgery affecting drug absorption, open biopsy, severe traumatic injury, wound unhealed or did not recover from major surgery within 1 month before the trial;
4. Before the first administration, patients have used strong CYP3A inhibitors (such as itraconazole, telithromycin, clarithromycin, ritonavir, etc.) or medium CYP3A inhibitors (such as ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil, etc.); Patients who had used strong CYP3A inducers (e.g., phenobarbide, enzyluamide, phenytoin, rifampicin, rifambutin, rifapentine, carbamazepine, nevirapine and St. John's herb) or medium CYP3A inducers (e.g., Bosentan, efavirenz, modafinil, etc.) and did not reach 3 elimination half-lives;
5. Pregnant or lactating women or subjects who cannot use contraception as required;
6. Those who have special requirements on diet and cannot accept uniform diet;
7. As judged by the researcher, there are other circumstances that are not suitable for the researcher.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-12-24 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free-Survival | 2 years
  The length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse

SECONDARY OUTCOMES:
Objective remission rate | 2 years
  It refers to the proportion of patients (mainly solid tumors) whose tumor has shrunk to a certain extent and remained there for a certain period of time, including Complete Response (CR) and Partial Response (PR).
Overall Survival | 2 years
  Time from randomization to death from any cause (for subjects who have been lost to follow-up prior to death, the time of death is usually calculated as the time of last follow-up)
Adverse event Adverse event | 2 years
  It refers to all adverse medical events that occur after a subject receives an investigational drug, which may be manifested as symptoms, signs, diseases, or abnormalities in laboratory tests, but may not necessarily be causally related to the investigational drug

CONTACTS AND LOCATIONS:
Overall Officials: Haiyan Liu, Principal Investigator — The Second Affiliated Hospital of Shandong First Medical University
Locations (1):
- The Second Affiliated Hospital of Shandong First Medical University, Tai’an, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Domchek SM, Aghajanian C, Shapira-Frommer R, Schmutzler RK, Audeh MW, Friedlander M, Balmana J, Mitchell G, Fried G, Stemmer SM, Hubert A, Rosengarten O, Loman N, Robertson JD, Mann H, Kaufman B. Efficacy and safety of olaparib monotherapy in germline BRCA1/2 mutation carriers with advanced ovarian cancer and three or more lines of prior therapy. Gynecol Oncol. 2016 Feb;140(2):199-203. doi: 10.1016/j.ygyno.2015.12.020. Epub 2015 Dec 23. PMID 26723501
- [Background] Moore KN, Secord AA, Geller MA, Miller DS, Cloven N, Fleming GF, Wahner Hendrickson AE, Azodi M, DiSilvestro P, Oza AM, Cristea M, Berek JS, Chan JK, Rimel BJ, Matei DE, Li Y, Sun K, Luptakova K, Matulonis UA, Monk BJ. Niraparib monotherapy for late-line treatment of ovarian cancer (QUADRA): a multicentre, open-label, single-arm, phase 2 trial. Lancet Oncol. 2019 May;20(5):636-648. doi: 10.1016/S1470-2045(19)30029-4. Epub 2019 Apr 1. PMID 30948273
- [Background] Mellinghoff IK, Chang SM, Jaeckle KA, van den Bent M. Isocitrate Dehydrogenase Mutant Grade II and III Glial Neoplasms. Hematol Oncol Clin North Am. 2022 Feb;36(1):95-111. doi: 10.1016/j.hoc.2021.08.008. Epub 2021 Oct 25. PMID 34711457
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961